CLINICAL TRIAL: NCT05272397
Title: The Interaction of Cognitive Control Mechanisms and Language Processing: An Investigation With Methylphenidate
Brief Title: Language & Cognitive Control
Acronym: LCCMPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donders Centre for Cognitive Neuroimaging (Other)
Collaborators: Max Planck Institute for Psycholinguistics (Unknown); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL69700.091.19
Record Dates: First submitted 2022-02-07; First posted 2022-03-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-02

CONDITIONS: Language; Methylphenidate of Undetermined Intent
Keywords: Cognitive Control; Language Processing; Reading; Methylphenidate; Catecholaminergic Neurotransmitters
MeSH Terms: conditions — Language | interventions — Methylphenidate; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug Session (Active Comparator): In this arm of the study participants receive the drug (Methylphenidate - 20mg), administered prior to completion of the primary and secondary tasks for the study.
  Electroencephalography (EEG) is measured for the duration of the primary and secondary tasks. Participants complete both arms of the study, and the order in which participants are assigned to this and the other arm of the study is randomized.
  Interventions: Drug: Methylphenidate 20 Mg Oral Tablet; Behavioral: Language Task; Behavioral: Rest Recording; Behavioral: Go/No-Go Task; Behavioral: Processing Speed
- Placebo Session (Placebo Comparator): In this arm of the study participants receive the a placebo, administered prior to completion of the primary and secondary tasks for the study.
  Electroencephalography (EEG) is measured for the duration of the primary and secondary tasks. Participants complete both arms of the study, and the order in which participants are assigned to this and the other arm of the study is randomized.
  Interventions: Drug: Placebo; Behavioral: Language Task; Behavioral: Rest Recording; Behavioral: Go/No-Go Task; Behavioral: Processing Speed
- Intake Session (Other): In this arm of the study participants are screened for suitability to participate in the experiment based on specified inclusion and exclusion criteria. They also complete some baseline tasks to assess working memory capacity, impulsiveness, and subjective mood.
  Interventions: Behavioral: Operation Span; Behavioral: Reading Span; Behavioral: Barratt Impulsiveness Scale

INTERVENTIONS:
Drug: Methylphenidate 20 Mg Oral Tablet — 20mg methylphenidate or placebo capsule - one per session (counterbalanced) approximately 1 week apart
  Arms: Drug Session
Drug: Placebo — 20mg methylphenidate or placebo capsule - one per session (counterbalanced) approximately 1 week apart
  Arms: Placebo Session
Behavioral: Language Task — The core part of the experiment is the language task, in which the aim is to investigate two critical aspects of language processing: semantic and syntactic processing. In this task, participants will be asked to read a list of sentences.
  Arms: Drug Session; Placebo Session
Behavioral: Rest Recording — Brain activity in the EEG is recorded at rest with eyes open and eyes closed to obtain baseline measures of alpha power as a proxy for attention and control under conditions of drug and placebo.
  Arms: Drug Session; Placebo Session
Behavioral: Go/No-Go Task — A Go/No-Go task will be implemented in the study design to investigate the functional properties of spatial selective attention and response inhibition. An adapted cued Go/No-Go paradigm from Randall & Smith (2011) will be employed.
  Arms: Drug Session; Placebo Session
Behavioral: Processing Speed — A speeded button response task will be included to measure participants' general processing speed. In this task, participants will be instructed to respond to a simple shape presented in the centre of the screen as fast and accurately as possible through pressing a corresponding button.
  Arms: Drug Session; Placebo Session
Behavioral: Operation Span — In the operation span task, participants are instructed to solve math operations (e.g., (1*2) +1=?) as soon as possible and then remember a single letter. This to-be-remembered letter is followed by either another math-word combination or a recall screen, which will show up at the end of each set. When the recall screen is presented, participants have to recall all the letters in the correct order they were presented. The experimental trials contain three sets at each set size (i.e., the number of math-word pairs), with set sizes ranging from 3 to 7 items. This results in a total of 75 sets with 75 letters and 75 math problems. The order of set sizes is random for each participant. Participants' operation span will be evaluated by the total number of letters recalled in the correct serial position regardless of whether the entire trial was recalled correctly.
  Arms: Intake Session
Behavioral: Reading Span — Participants are instructed to judge whether a presented sentence makes sense or not. After each sentence, a to-be-remembered letter will be shown on the screen, which is followed by either another sentence-word combination or the final recall screen. The set size ranges from 3 to 7 items. At the end of each set of sentences, participants will be required to recall all the letters in the current set in order. There will be a total of 75 letters and 75 sentence judgements. The order of the set sizes will be at random for each participant. Participants' performance will be evaluated by calculating the total number of correctly recalled letter sets.
  Arms: Intake Session
Behavioral: Barratt Impulsiveness Scale — The Barratt impulsiveness scale (BIS-11) will be used in the experiment to measure participants' trait impulsivity. Participants will be required to rate themselves on 30 items that are related to attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness.
  Arms: Intake Session

SUMMARY:
Catecholamine (CA) neurotransmitters, such as dopamine (DA) and noradrenaline (NA), have long been implicated playing a critical role in cognitive functions, such as working memory (WM), inhibition, learning, and decision making. Recent evidence from neurodegenerative patients and the healthy population suggested that CA also influences language processing. However, the question of what kind of influence that CA might exert on language is still open. Some previous studies have shown that CA can enhance semantic processing. In a recent study it was observed that CA agonists (i.e., methylphenidate) enhance participant's sensitivity to semantically incongruent information even when language processing was actually goal-irrelevant. On the other hand, the processing of semantically congruent information was enhanced while language processing was the goal. Moreover, consistent with some previous findings that there is a relation between participants' baseline characteristics and MPH effects, it was observed that participants with lower WM capacity benefited more from receiving methylphenidate. These results shed light on the relation between CA and language processing, but also lead to further questions, such as whether the interaction between CA and semantic processing is language-specific or mediated by the relation between CA and more general cognitive functions (e.g., WM, inhibition), and whether CA also has an influence on other aspects of language processing, such as syntactic processing. The present study aimed to further investigate the nature of the relation between CA and language processing by administrating methylphenidate (MPH) to healthy participants. MPH is an indirect CA agonist, which is the most commonly prescribed drug for attention deficit/hyperactivity disorder (ADHD). Previous studies have shown that MPH can efficiently increase the extracellular levels of CA in the brain by blocking their reuptake.

Objective: The primary objectives are: 1) to further investigate the effect of CA on semantic processing. The study plans to examine whether MPH interacts with processing of sentence context constraints via its influence on cognitive control operations. 2) To investigate the effects of MPH on syntactic processing. More specifically, the study is interested in whether MPH has an influence on revising syntactically temporarily ambiguous sentences.

A secondary objective is to further examine the relation between MPH effects and the baseline characteristics of individual participants.

Study design: This study will use a within-subject, double-blind, placebo-controlled, randomized, crossover design.

Study population: Approximately 40 healthy native Dutch speakers between 18 and 45 years old will be recruited. All subjects will have to complete one screening session and two separate testing sessions within three different days at the Donders Centre for Cognitive Neuroimaging (DCCN).

Intervention: Participants will either orally receive a 20mg methylphenidate or placebo capsule in each of the two testing sessions. Methylphenidate has been approved for clinical use in the Netherlands and the drug can be administered safely without any relevant risk of serious adverse events.

Main study parameters: Primary study parameters will include sentence comprehension capacity, attention and processing speed. In addition, several other measures will be included to monitor participants' baseline characteristics (e.g. working memory capacity, vocabulary size) and the general modulation effects of MPH (e.g. heart rate, blood pressure, subjective feeling).

Hypotheses:

Based on the previous finding that methylphenidate improves cognitive stability while it impairs flexible updating, the hypothesis is that methylphenidate will hinder participants' performance in resolving syntactic ambiguity, which requires an immediate updating and revising of an initial interpretation. This should be reflected in event-related potential (ERP) measures related to revision, namely the P600 effect is predicted to be reduced in the drug condition compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Native Dutch speakers
* Right-handed

Exclusion Criteria:

* Current (or history of) psychiatric disorder (e.g., psychosis, mania, severe depressive disorder)
* Current (or history of) neurological disorder (e.g. m. Parkinson, epilepsy)
* Current (or history of) endocrine / metabolic disorder
* Current (or history of) cardiac or vascular disorder
* Current (or history of) blood illness (e.g. severe anaemia, porphyria)
* Current (or history of) stomach or gastrointestinal tract disease
* History of autonomic failure (e.g., vasovagal reflex syncope)
* Experience of irregular sleep-wake rhythm
* Current (or history of) obstructive respiratory disease
* Current (or history of) clinically significant renal or hepatic disease
* (Recent treatment of) glaucoma
* Current (or history of) drug addiction (e.g. opiate, (meth)amphetamine, lysergic acid diethylamide, cocaine, solvents or barbiturate) or alcohol dependence
* One first degree or two or more second degree family members with a recent treatment of sudden death or ventricular arrhythmia
* Problems swallowing or problems with the oesophagus
* Frequent experience of headrush (vertigo)
* Current experience of an acute serious infection
* First degree family member with schizophrenia or bipolar disorder
* Abnormal hearing or (uncorrected) vision
* Use of psychotropic medication or recreational drugs weekly or more over a period of more than three months in the last 6 months
* Cannabis usage for the last 6 months
* Strong smoking behaviour starting at more than 1 package of cigarettes per week
* Hypersensitivity for e.g. beta blockers or methylphenidate
* Uncontrolled hypertension, defined as diastolic blood pressure at rest >95 mmHg or systolic blood pressure at rest >180 mmHg
* Irregular sleep/wake rhythm (e.g. regular nightshifts or cross timeline travel)
* Possible pregnancy or breastfeeding/ inadequate anticonception (for women)
* Lactose intolerance (because the placebo pill will be a lactose product)
* Language related disabilities (e.g. dyslexia, stuttering)
* Daily intense physical training

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Language Task ERP Drug Session | First or second testing session depending on which session corresponds to the session where the drug was administered.
  This measure will assess the P600 ERP effect (amplitude difference between correct and syntactic ambiguity conditions) just after the target word in the sentences being read.
Language Task ERP Placebo Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  This measure will assess the P600 ERP effect (amplitude difference between correct and syntactic ambiguity conditions) just after the target word in the sentences being read.
Language Task Alpha Power Drug Session | First or second testing session depending on which session corresponds to the session where the drug was administered.
  This measure will assess the alpha power effect (relative power difference between high and low sentence constraint conditions in the alpha frequency band, 8-12 Hz) just before the target word in the sentences being read.
Language Task Alpha Power Placebo Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  This measure will assess the alpha power effect (relative power difference between high and low sentence constraint conditions in the alpha frequency band, 8-12 Hz) just before the target word in the sentences being read.

SECONDARY OUTCOMES:
Default Mode Alpha Power Drug Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  This measure will assess alpha power (8-12 Hz) at rest (relative difference between alpha power measured over the duration of the eyes open to that measured over the duration of the eyes closed recordings).
Default Mode Alpha Power Placebo Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  This measure will assess alpha power (8-12 Hz) at rest (relative difference between alpha power measured over the duration of the eyes open to that measured over the duration of the eyes closed recordings).
Go-NoGo Task Alpha Power Drug Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  This measure will assess alpha power (8-12 Hz) at response and no-response cues to obtain a measure of attentional control.
Go-NoGo Task Alpha Power Placebo Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  This measure will assess alpha power (8-12 Hz) at response and no-response cues to obtain a measure of attentional control.

OTHER OUTCOMES:
Peabody Picture Vocabulary Test | First testing session.
  The Peabody Picture Vocabulary Test (PPVT) is used to measure vocabulary size. Raw scores are converted to standardized scores based on normative age-matched data (μ = 100; σ = 15). A higher score indicates better performance.
General Processing Speed Drug Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  Participants respond as fast as possible via button-press to a shape presented on the screen. Reaction time (RT) and accuracy are combined to obtain a single measure of performance, with faster RTs indicating better performance.
General Processing Speed Placebo Session | First or second testing session depending on which session corresponds to the session where the placebo was administered.
  Participants respond as fast as possible via button-press to a shape presented on the screen. Reaction time (RT) and accuracy are combined to obtain a single measure of performance, with faster RTs indicating better performance.
Barratt Impulsiveness Scale | Intake Session, 1-4 weeks prior to the intervention sessions
  The Barrat Impulsiveness Scale (BIS) is used to assess the trait of impulsivity. Individual responses are scored on a 4-point scale (Rarely/Never = 1; Occasionally = 2; Often = 3; Almost always/Always = 4) and higher scores correspond to greater impulsivity.
Reading Span Task | Intake Session, 1-4 weeks prior to the intervention sessions
  Participants are required to memorize letters presented between sentences that have to be read. The outcome measure is the number of letters correctly recalled in the correct order in a subsequent memory test. Set sizes range from 3-7 letters before memory is tested. This provides a measure of working memory capacity. More letters recalled indicates better working memory performance.
Operation Span Task | Intake Session, 1-4 weeks prior to the intervention sessions
  Participants are required to memorize letters presented between math operations that have to be solved as quickly as possible. The outcome measure is the number of letters correctly recalled in the correct order in a subsequent memory test. Set sizes range from 3-7 letters before memory is tested. This provides a measure of working memory capacity. More letters recalled indicates better working memory performance.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hagoort, PhD, Principal Investigator — Donders Centre for Cognitive Neuroimaging
Locations (1):
- Donders Institute for Brain, Cognition and Behaviour, Centre for Cognitive Neuroimaging, Nijmegen, Gelderland, Netherlands